CLINICAL TRIAL: NCT05041036
Title: Individual Patient Compassionate Use of Nirogacestat
Status: Available | Type: Expanded Access
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIR-DT-701
Record Dates: First submitted 2021-09-07; First posted 2021-09-10 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Desmoid Tumor; NOTCH Gene Mutation Positive Tumors
Keywords: desmoid tumor; aggressive fibromatosis; desmoid fibromatosis; Notch-positive tumors
MeSH Terms: conditions — Desmoid Tumors | interventions — nirogacestat

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Nirogacestat (Gamma Secretase Inhibitor) — Patients will receive nirogacestat tablets to be taken orally.

SUMMARY:
This program is being offered on a patient by patient basis and will require company, Institutional Review Board/Independent Ethics Committee, and applicable competent authority approval.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a serious, debilitating or life-threatening medical condition that cannot be treated satisfactorily with an authorized medicinal product or other available standard treatment options, or all other treatment options have been exhausted.
* Patient does not qualify to participate in an ongoing clinical trial.

Sex: All
Age Groups: Child, Adult, Older Adult